CLINICAL TRIAL: NCT06389578
Title: A Phase 1b, Open-label, Multicenter Trial to Evaluate the Pharmacokinetics, Safety, and Tolerability of Two Formulations of a Single Subcutaneous Dose of Teprotumumab Followed by Multiple Intravenous Doses of TEPEZZA in Participants With Thyroid Eye Disease
Brief Title: A Study of TEPEZZA® Treatment in Participants With Thyroid Eye Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-TEP-103
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Thyroid Eye Disease
Keywords: Thyroid Eye Disease; TEPEZZA; Teprotumumab
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive a single dose of lyophilized teprotumumab by subcutaneous (SC) administration on Day 1 followed by intravenous (IV) infusions of teprotumumab at the approved dosing regimen.
  Interventions: Drug: Teprotumumab
- Cohort 2 (Experimental): Participants will receive a single high concentration formulation teprotumumab by SC administration on Day 1 followed by IV infusions of teprotumumab at the approved dosing regimen.
  Interventions: Drug: Teprotumumab

INTERVENTIONS:
Drug: Teprotumumab — SC administration and IV infusion
  Other Names: Tepezza

SUMMARY:
The main goal of this study is to learn how teprotumumab will be processed in the body (Pharmacokinetics) subcutaneously and whether it is safe and tolerable after administration into adult patients with thyroid eye disease.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter trial to assess the PK, safety, and tolerability of a single SC dose of lyophilized teprotumumab and high concentration formulation teprotumumab in participants with thyroid eye disease. Approximately 6 participants (in Cohort 1) and approximately 10 participants (in Cohort 2) who meet the trial eligibility criteria will be enrolled in a 1:1 ratio.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Thyroid eye disease (not sight-threatening but has an appreciable impact on daily life), usually associated with one or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, proptosis, and/or inconstant or constant diplopia.
2. Proptosis ≥ 3 mm increase from the participant's baseline (prior to diagnosis of TED), as estimated by treating physician and/or proptosis ≥ 3 mm above normal for race and gender.
3. Participant must be euthyroid with baseline disease under control or have mild hypo- or hyperthyroidism at Screening. Every effort should be made to correct the mild hypo or hyperthyroidism promptly and to maintain the euthyroid state for the full duration of the trial.
4. Does not require immediate surgical ophthalmological intervention.
5. Participants with diabetes must have HbA1c ≤ 8.0% at Screening.

Exclusion Criteria:

1. Decreased best-corrected visual acuity due to optic neuropathy within the last 6 months.
2. Corneal decompensation unresponsive to medical management in the study eye.
3. Decrease in proptosis of ≥ 2 mm in the study eye between Screening and Baseline.
4. Alanine aminotransferase or aspartate aminotransferase > 3x the upper limit of normal or estimated glomerular filtration rate ≤ 30 mL/min/1.73 m2 at Screening.
5. Use of any steroid (IV, oral, steroid eye drops) for the treatment of TED or other conditions within 3 weeks prior to Screening. Steroids cannot be initiated during the trial. Exceptions include topical and inhaled steroids and steroids used to treat infusion reactions.
6. Any treatment with rituximab, tocilizumab, or any other non-steroid immunosuppressive agent within 90 days prior to the first injection of investigational product on Day 1.
7. Any previous treatment with HZN-001 or TEPEZZA (teprotumumab-trbw), including previous enrollment in this trial or participation in a prior TEPEZZA trial.
8. Treatment with any mAb within 3 months prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Curve (AUC) of Teprotumumab | Pre dose through Week 6
  AUC will be evaluated from the collected PK samples.
PK: Maximum Serum Concentration (Cmax) of Teprotumumab | Pre dose through Week 6
  Cmax will be evaluated from the collected PK samples.
Number of Participants With Adverse Events (AE) | Up to Week 6
  An AE is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Bascom Palmer Eye Institute - University of Miami, Miami, Florida
  - Barnes Jewish Hospital Washington University, St Louis, Missouri
  - Neuro-Eye Clinical Trials, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing